CLINICAL TRIAL: NCT01167647
Title: The Role of Routine Bacterial Culture Including Tuberculosis During
Brief Title: The Role of Routine Bacterial Culture Including Tuberculosis During Bronchoscopy: A Prospective Study
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MMC10-087-10.CTIL
Record Dates: First submitted 2010-07-21; First posted 2010-07-22 (Estimated); Last update posted 2013-03-06 (Estimated); Status verified 2012-03

CONDITIONS: Tuberculosis
Keywords: Tuberculosis, culture, bronchoscopy
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- bronchoscopy patients

SUMMARY:
Many centers routinely culture bronchoscopy samples for bacteria and mycobacteria even when infections including tuberculosis (TB) are not strongly suspected. However, the value of this practice has been poorly defined.

DETAILED DESCRIPTION:
Many centers routinely culture bronchoscopy samples for bacteria and mycobacteria even when infections including tuberculosis (TB) are not strongly suspected. However, the value of this practice has been poorly defined. Unnecessary bronchial cultures of bacteria may lead to over treatment in patients without clinical evidence of infections and may increase the drug resistant strains.

In areas with a high prevalence of TB, routine bronchial cultures may detect clinically unsuspected TB in an appreciable proportion of cases. However, in population with a low prevalence of TB, routine culture of bronchial aspirates may incur an unnecessary expanse and may lead to over diagnosis and over treatment of patients with non pathogenic atypical mycobacteria detected by acid-fast bacillus strains.

ELIGIBILITY:
Inclusion Criteria:

1. patients who will undergo a bronchoscopy examination at pulmonary department in Meir Medical Center
2. patients who will sign on informed consent. -

Exclusion Criteria:

* 1)age under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who will undergo a bronchoscopy examination at pulmonary department in Meir Medical Center and will sign on informed consent.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2010-07; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
number of positive tuberculosis culture | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: David Shitrit, MD, Principal Investigator — Meir Medical Center
Locations (2):
- Israel (2):
  - Pulmonary department, Meir Medical Center, Kfar Saba, Israel
  - Pulmonary department, Meir Medical Center, Kfar Saba

REFERENCES:
- [Derived] Talker O, Matveychuk A, Guber A, Mandelbaum-Livnat MM, Varsano S, Shitrit D. Is routine bronchoscopic culture indicated in areas with low tuberculosis prevalence? Int J Tuberc Lung Dis. 2013 Aug;17(8):1100-3. doi: 10.5588/ijtld.12.0997. PMID 23827036